CLINICAL TRIAL: NCT03519399
Title: Investigation of the Effect of Elevated Serum Bile Acids in Intrahepatic Cholestasis of Pregnancy (ICP) on the Fetal Cardiac Rhythm and on Myometrial Contractility: a Prospective Case-control Pilot Study
Brief Title: Bile Acid Effects in Fetal Arrhythmia Study
Acronym: BEATS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: RJ115/N071
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Cholestasis of Pregnancy; Intrahepatic Cholestasis of Pregnancy; Obstetric Cholestasis
Keywords: Bile Acids, Fetal ECG, Stillbirth,
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Stillbirth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal sera samples collected at recruitment. Maternal sera and umbilical cord blood sera collected following the delivery of the fetus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases and Controls: Cases - Pregnant women with ICP defined as pruritus in pregnancy in association with raised serum bile acids (using hospital threshold for diagnosis), and in the absence of an alternative cause.
  Controls - Pregnant women not affected by ICP, or other liver, cardiac or hypertensive disorders.
  Interventions: Device: Monica AN24

INTERVENTIONS:
Device: Monica AN24 — Monica AN24 will be used to record maternal and fetal ECGs. The Zephyr will be used to determine maternal lie.
  Other Names: Zephyr

SUMMARY:
Intrahepatic cholestasis of pregnancy (ICP) is a liver disorder of pregnancy that typically presents in late pregnancy with generalised itching. ICP is associated with an increased risk of pregnancy complications, including premature labour, fetal distress, and stillbirth. Models of the fetal heart (using cells from rodents) have shown that high bile acids levels cause an abnormal heart rhythm (arrhythmia), which may be the cause of stillbirth. High levels of bile acids also cause preterm labour in animal models.

This pilot study aims to assess whether severe ICP, defined as maternal serum bile acid levels ≥40μmol/L, is associated with abnormal fetal heart rhythms and abnormal myometrial contractility, which may lead to preterm birth.

Fetal heart rhythms and myometrial contractility will be recorded using a portable electrocardiogram (ECG) device, the Monica AN24. This monitors the fetal heart and myometrial activity via stickers applied to the mother's abdomen. It also records the maternal ECG. It will also study women with uncomplicated pregnancy, in order to make comparisons.

The importance of maternal position during sleep has also more recently been established, with some studies demonstrating an association between the risk of stillbirth and the position the mother was sleeping in. Work by Stone et al published this year has shown that the maternal sleep position has a significant impact on the fetal sleep state and fetal heart rate, (in particular something called the fetal RMSSD value). The researchers therefore wish to identify any potential correlation between fetal heart arrhythmia and maternal sleep position. To do this they will use a Zephyr BioPatchTM which provides a clear indication of whether the patient was in left lateral, right lateral or supine position.

DETAILED DESCRIPTION:
Intrahepatic cholestasis of pregnancy (ICP) also known as obstetric cholestasis (OC) is a liver disorder unique to pregnancy that affects 0.5-1% of women in the UK. It typically presents in the third trimester of pregnancy with pruritus that can affect any part of the body, but is most commonly experienced on the palms and soles. Biochemically, it is characterised by liver dysfunction with raised serum bile acids, and clinically, by a significantly increased incidence of fetal complications, including spontaneous preterm labour, fetal distress, meconium staining of the amniotic fluid and sudden fetal death

The aetiology of ICP is complex and incompletely understood although the maternal disease is likely to be caused by interaction between sex hormone metabolites and bile acids in genetically susceptible women . To date, genetic variation in several biliary transporters have been identified that predispose women to the disease. The aetiology of the adverse perinatal outcomes is also not fully understood.

ICP is associated with an increased risk of adverse perinatal outcomes, including spontaneous preterm delivery, meconium staining of the amniotic fluid, admission to the neonatal unit and sudden intrauterine death. As with the maternal disease, the aetiology for the perinatal complications is not fully understood, but evidence from animal and in vitro studies suggests a role for bile acids. This hypothesis is supported by the finding that the risk of adverse perinatal outcomes is directly associated with the level of maternal serum bile acids, and specifically with maternal serum bile acids exceeding 40 μmol /L, i.e. severe ICP.

Of the adverse perinatal outcomes associated with ICP, the most severe is sudden intrauterine death, which is reported to affect between 2 and 4% of ICP pregnancies. The mechanism for fetal demise is unclear, but is appears to be a sudden event as there are several case reports of normal fetal movements and CTG recordings in the hours preceding fetal demise. Furthermore, at post-mortem there is typically no evidence of preceding uteroplacental insufficiency, and the babies are appropriately grown. One possible explanation for the sudden intrauterine death is an acute cardiac arrhythmia leading to fetal cardiac arrest. This hypothesis is supported by evidence from in vitro studies of cultured neonatal rat cardiomyocytes which demonstrate the development of arrhythmias following the addition of bile acids to the culture (Williamson et al., 2001). Further studies have shown that this effect is dose dependent and reversed by the addition of ursodeoxycholic acid (UDCA), the drug commonly used to treat ICP. However, there are very few case reports in the literature of fetal heart abnormalities in women with ICP, but studies have reported bradycardias, tachycardias and atrial flutter. Prolongation of the PR interval in the fetal echocardiogram has also been reported; this clinical feature has been known to predispose the heart to arrhythmias. A recent study using the same technique has also reported fetal diastolic dysfunction in patients with severe ICP. Given the paucity of human clinical data regarding the fetal heart rhythm in ICP, the researchers propose to undertake this study to investigate whether ICP is associated with fetal arrhythmias and the influence of bile acid levels on fetal heart rhythm. In parallel they will evaluate whether there is fetal ventricular dysfunction.

Recent studies have shown that maternal lie has an association with stillbirth; an increased risk of stillbirth was observed when women slept in a supine or right lateral position. Stone et al published data from a study where the Monica AN24, a transabdominal fetal electrocardiogram (fECG) monitor, was used on mothers lying in supine, left and right lateral positions. They found that the fetal short-term heart rate variability (RMSSD) changed depending on the position the mother was lying in. Unpublished data also using the Monica AN24 has demonstrated an association between maternal lie and maternal RMSSD (Fifer et al, personal communication). As the RMSSD is one of the principal measures the research team will be using to detect arrhythmogenic activity, analysis will include the detection of maternal lie in order to accurately determine short-term heart rate variability.

There is limited evidence that the maternal heart is affected by ICP to cause maternal rhythm disturbance, although there is one report of prolonged maternal QT interval. The fetal heart develops in an environment of relative hypoxia and this is associated with the transformation of human fetal cardiac fibroblasts into myofibroblasts, which subsequently disappear post-natally. Myofibroblasts may re-appear in the diseased adult heart during the process of remodelling following infarction, and have been shown to act as an arrhythmogenic focus in these circumstances. Interestingly, in vitro data have demonstrated that the myofibroblasts also act as the arrhythmogenic focus in bile acid induced arrhythmia in the neonatal heart. UDCA has also been demonstrated to protect against bile acid-induced arrhythmias in myofibroblasts.

ICP is also associated with an increased risk of spontaneous preterm labour. Again, the reasons for this are unclear, but evidence from animal studies suggests that bile acids may be involved. Bile acid infusions cause spontaneous preterm labour in sheep and in vitro studies have shown that they increase the sensitivity of the myometrium to the hormone oxytocin which is central to the process of labour. Human data regarding myometrial contractility are lacking. As a secondary aim of this study, the research team also propose to investigate whether ICP is associated with abnormal myometrial contractility.

Data regarding fetal cardiac rhythms and myometrial contractility collected from women with ICP will be compared to data collected from women with uncomplicated pregnancy. The inclusion of women with uncomplicated pregnancies will ensure that any variation identified in the fetal cardiac rhythms or myometrial contractility in women with ICP is attributable to the condition, rather than a variant of normal. The parallel recording of the maternal ECG in both women with ICP and women with uncomplicated pregnancy will enable the research team to ensure that any abnormal fetal cardiac rhythms are not due to an inherited arrhythmia.

Fetal and maternal ECG, and myometrial contractility data will be collected using the Monica AN24 device. This is a small wearable monitor that continuously records maternal and fetal ECG's, and myometrial activity data via electrodes placed on the maternal abdomen. Maternal lie will be detected using the Zephyr BioPatchTM. This wearable monitor is much smaller than the Monica AN24 and also functions via adhesive electrodes. It is placed at the base of the breastbone of the participant.

ELIGIBILITY:
Inclusion Criteria:

* CASES - Pregnant women with ICP defined as pruritus in pregnancy in association with raised serum bile acids (using hospital threshold for diagnosis), and in the absence of an alternative cause.
* CONTROLS - Pregnant women not affected by ICP, or other liver, cardiac or hypertensive disorders.
* Pregnant women who are willing and able to give consent.
* Pregnant women ≥ 18 years of age.

Exclusion Criteria:

* Non-pregnant women.
* Pregnant women with medical disorders that can cause liver impairment in pregnancy e.g. pre-eclampsia, acute fatty liver of pregnancy, diabetes mellitus.
* Pregnant women with a history of pre-existing liver or cardiac
* Pregnant women with current hypertensive disease (this would include women taking drugs such as methyldopa, labetolol, atenolol, bisoprolol, nifedipine, amlodipine)
* Pregnant women who are expecting more than one baby.
* Pregnant women with blood-borne viruses e.g. HIV and hepatitis.
* Women ≤ 18 years of age.
* Pregnant women expecting a baby with a structural heart abnormality identified
* Women unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible women will be identified via the antenatal services at participating hospitals, and via ICP support (www.icpsupport.org).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-02-27 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of the influence of maternal bile acids levels on fetal ECG | Up to 24 hours (overnight recording at home)
  To investigate the influence of maternal serum bile acid levels on the fetal ECG in women with ICP and women with uncomplicated pregnancy.

SECONDARY OUTCOMES:
Measurement of the influence of fetal bile acids levels on fetal ECG | Up to 24 hours (overnight recording at home)
  To investigate associations between fetal bile acid levels and the fetal ECG in women with ICP and women with uncomplicated pregnancy
Measurement of the influence of maternal bile acids levels on myometrial contractility | Up to 24 hours (overnight recording at home)
  To investigate associations between maternal serum bile acid levels and myometrial contractility in women with ICP and women with uncomplicated pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Williamson, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - St Thomas' Hospital, London
  - Queen Charlotte's & Chelsea Hospital, London